CLINICAL TRIAL: NCT00869349
Title: Brigham Rheumatoid Arthritis Sequential Study B.R.A.S.S.
Brief Title: Living Well With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Nancy Shadick, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2002-P-001762
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; IFS; psychosocial; social support
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IFS Intervention Group (Experimental)
  Interventions: Behavioral: IFS
- Education Group (Active Comparator)
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: IFS — The program will begin with a half day orientation to meet the trained professional coaches and other patients enrolled in the program. Following the orientation there will be group meetings of 8-10 RA patients every other week for twelve weeks with one of the trained coaches. In the weeks patients do not meet with the group, patients will have individual coaching sessions. The group meetings will last approximately 90 minutes and the individual meetings will last 50 minutes. A maintenance program will follow with bimonthly coaching sessions and a group meeting once a month over the next six months.
  Three, six and nine months after the beginning of the program, patients will return to the hospital to complete the same research questionnaire and physical examination they received at baseline.
  Arms: IFS Intervention Group
Other: Education — The intervention for the controls includes an initial meeting with a health professional. Once a month for 9 months, patients will received educational material and a follow-up phone call to ask if the patient received the information and to answer any questions about the material.
  Arms: Education Group

SUMMARY:
The purpose of the Living Well with RA program is to perform a proof-of-concept study and evaluate the efficacy of an Internal Family Systems-based psychotherapeutic intervention improve Rheumatoid Arthritis subjects' disease activity, independence and other health outcomes. This study will also assess the efficacy of an IFS-based program in improving RA subjects' mental health symptoms. We hypothesize that the IFS model will improve RA subjects self-management of their disease and subsequently their health outcomes will improve as well as compared to a group focusing on arthritis education.

DETAILED DESCRIPTION:
Subjects will be selected from the Brigham & Women's Hospital Arthritis Center and include those enrolled in the BRASS study and then once recruited randomly assigned to either the IFS intervention group or the education group. Both the IFS intervention and education group will participate in their respective programs simultaneously over 9 months.

Subject reported measures:

Incorporated into the questionnaires are several subject-reported measures, including: The Self-Compassion Scale, Beck Depression Index (BDI-II), SF-12 Health Survey, State-Trait Anxiety Inventory (STAI), RA Disease Activity Index (RADAI), and Arthritis Self-Efficacy Scale. These measures report emotional states, degree and location of arthritis pain, and how that pain affects their daily lives. A monthly encounter form will also be completed by the subject.

Physician measures:

The physicians who will be monitoring subject health are blind to the study and complete the same measures for subjects in both the IFS intervention and education groups. They will complete a joint count, Global Assessment of health, duration of morning stiffness and ACR functional status.

Laboratory testing:

Subjects will give blood at the beginning, 3, 6 and 9-month points of the program. This sample will be laboratory-tested for C-reactive protein.

Data collection schedule:

Subjects will complete a questionnaire at baseline, then at 3, 6 and 9 months. They will give blood samples and undergo a routine physical examination, focusing on their joints at the initial meeting, again at 3, 6, and 9 months into the study.

ELIGIBILITY:
Inclusion Criteria:

* Active RA symptoms
* Member of the BRASS registry at the Brigham and Women's Arthritis Clinic
* Ability to attend group and individual sessions consistently

Exclusion Criteria:

* RA has been in remission for one year
* Subjects who are currently enrolled in the Arthritis Foundation Self- Management course or any similar type of course

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Shadick, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Achterberg J, McGraw P, Lawlis GF. Rheumatoid arthritis: a study of relaxation and temperature biofeedback training as an adjunctive therapy. Biofeedback Self Regul. 1981 Jun;6(2):207-23. doi: 10.1007/BF00998870. PMID 7020777
- [Background] Astin JA, Beckner W, Soeken K, Hochberg MC, Berman B. Psychological interventions for rheumatoid arthritis: a meta-analysis of randomized controlled trials. Arthritis Rheum. 2002 Jun 15;47(3):291-302. doi: 10.1002/art.10416. PMID 12115160
- [Background] Bradley LA, Young LD, Anderson KO, Turner RA, Agudelo CA, McDaniel LK, Pisko EJ, Semble EL, Morgan TM. Effects of psychological therapy on pain behavior of rheumatoid arthritis patients. Treatment outcome and six-month followup. Arthritis Rheum. 1987 Oct;30(10):1105-14. doi: 10.1002/art.1780301004. PMID 3314877
- [Background] Elenkov IJ, Chrousos GP. Stress hormones, proinflammatory and antiinflammatory cytokines, and autoimmunity. Ann N Y Acad Sci. 2002 Jun;966:290-303. doi: 10.1111/j.1749-6632.2002.tb04229.x. PMID 12114286
- [Background] Lorig K, Lubeck D, Kraines RG, Seleznick M, Holman HR. Outcomes of self-help education for patients with arthritis. Arthritis Rheum. 1985 Jun;28(6):680-5. doi: 10.1002/art.1780280612. PMID 4004977
- [Background] Lundgren S, Stenstrom CH. Muscle relaxation training and quality of life in rheumatoid arthritis. A randomized controlled clinical trial. Scand J Rheumatol. 1999;28(1):47-53. doi: 10.1080/03009749950155788. PMID 10092165
- [Background] O'Leary A, Shoor S, Lorig K, Holman HR. A cognitive-behavioral treatment for rheumatoid arthritis. Health Psychol. 1988;7(6):527-44. doi: 10.1037//0278-6133.7.6.527. PMID 3063517
- [Background] Parker, J. C., K.L. Smarr, S.P. Bucklew, R.C. Stucky-Ropp, J.E. Hewett (1995).
- [Background] Pradhan EK, Baumgarten M, Langenberg P, Handwerger B, Gilpin AK, Magyari T, Hochberg MC, Berman BM. Effect of Mindfulness-Based Stress Reduction in rheumatoid arthritis patients. Arthritis Rheum. 2007 Oct 15;57(7):1134-42. doi: 10.1002/art.23010. PMID 17907231
- [Background] Sharpe L, Sensky T, Timberlake N, Ryan B, Brewin CR, Allard S. A blind, randomized, controlled trial of cognitive-behavioural intervention for patients with recent onset rheumatoid arthritis: preventing psychological and physical morbidity. Pain. 2001 Jan;89(2-3):275-83. doi: 10.1016/s0304-3959(00)00379-1. PMID 11166484
- [Background] Shearn MA, Fireman BH. Stress management and mutual support groups in rheumatoid arthritis. Am J Med. 1985 May;78(5):771-5. doi: 10.1016/0002-9343(85)90282-7. PMID 3887910
- [Background] Smyth JM, Stone AA, Hurewitz A, Kaell A. Effects of writing about stressful experiences on symptom reduction in patients with asthma or rheumatoid arthritis: a randomized trial. JAMA. 1999 Apr 14;281(14):1304-9. doi: 10.1001/jama.281.14.1304. PMID 10208146
- [Background] Warsi A, LaValley MP, Wang PS, Avorn J, Solomon DH. Arthritis self-management education programs: a meta-analysis of the effect on pain and disability. Arthritis Rheum. 2003 Aug;48(8):2207-13. doi: 10.1002/art.11210. PMID 12905474
- [Background] Warsi A, Wang PS, LaValley MP, Avorn J, Solomon DH. Self-management education programs in chronic disease: a systematic review and methodological critique of the literature. Arch Intern Med. 2004 Aug 9-23;164(15):1641-9. doi: 10.1001/archinte.164.15.1641. PMID 15302634
- [Derived] Shadick NA, Sowell NF, Frits ML, Hoffman SM, Hartz SA, Booth FD, Sweezy M, Rogers PR, Dubin RL, Atkinson JC, Friedman AL, Augusto F, Iannaccone CK, Fossel AH, Quinn G, Cui J, Losina E, Schwartz RC. A randomized controlled trial of an internal family systems-based psychotherapeutic intervention on outcomes in rheumatoid arthritis: a proof-of-concept study. J Rheumatol. 2013 Nov;40(11):1831-41. doi: 10.3899/jrheum.121465. Epub 2013 Aug 15. PMID 23950186

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IFS Intervention Group | Education Group
Started | 39 | 40
Completed | 32 | 36
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IFS Intervention Group | Education Group | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.8) | 58.5 (12) | 58.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 38 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: RADAI Disease Activity Score
Description: Change in self-assessed disease activity from baseline to 21-months. Total RADAI score is 0-10 with 0 indicating no/low self-assessed disease activity and 10 indicating high self-assessed disease activity.
  Reference: Stucki G, Liang M, Stucki S, Bruhlmann P, Michel BA. A self-administered rheumatoid arthritis disease activity index (RADAI) for epidemiological research. Psychometric properties and correlation with parameters of disease activity. Arthritis Rheum. 38;795-98,1995
Time Frame: 21 months
Population: Data reported on per-protocol analysis. Sensitivity analysis was performed to evaluate robustness of analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IFS Intervention Group | Education Group
Number analyzed (Participants) | 32 | 36
units on a scale | -0.4 (1.1) | 0.1 (1.2)
Statistical Analysis 1: Comparison: IFS Intervention Group vs Education Group; Treatment effects are reported as mean between-group differences from baseline to 21 months using t-tests to determine the differential effect of the intervention versus the education group; Test type: Superiority or Other; p = 0.04, t-test, 2 sided — a priori threshold for statistical significance was <0.05; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to 0.0]

2. Secondary Outcome: Depression
Description: Change in the Beck Depression Scale from baseline to 21-months. The BDI-II (Reference: BDI- II Manual by Aaron T. Beck, Robert A. Steer, and Gregory K. Brown) is a 21-item scale for measuring negative attitudes about the future. Add up each of the items marked in the direction keyed for "hopelessness" to get a total score.
  Each of 21 items is summed to give single score for BDI-II.
  * There is 4-point scale ranging from 0 - 3. On 2 items (16, 18)
  * There are 7 options to indicate either increase or decrease of appetite and sleep. These are still scored 0 - 3 - answers are 0,1a,1b,2a,2b,3a,3b.
  * Cut score guidelines for the BDI-II are given with recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II.
    0 - 13 minimal 14 - 19 mild 20 - 28 moderate 29 - 63 severe
Time Frame: 21 months
Population: Data reported on per-protocol analysis. Sensitivity analysis was performed to evaluate robustness of analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IFS Intervention Group | Education Group
Number analyzed (Participants) | 32 | 36
units on a scale | -2.6 (4.3) | 0.6 (5.6)
Statistical Analysis 1: Comparison: IFS Intervention Group vs Education Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, t-test, 2 sided — a priori threshold for statistical significance was <0.05; Mean Difference (Net) = -3.2, 95% CI 2-sided [-5.6 to -0.8]

3. Secondary Outcome: Self-Compassion
Description: Change in the Neff Self Compassion scale from baseline to 21-months. This is a 26-item scale. The total self-compassion score ranges from 0 (no self-compassion) - 30 (high self-compassion). Reference: Neff, K.D. (2003). Development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250
Time Frame: 21 months
Population: Data reported on per-protocol analysis. Sensitivity analysis was performed to evaluate robustness of analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IFS Intervention Group | Education Group
Number analyzed (Participants) | 32 | 36
units on a scale | 1.8 (3.0) | 0 (2.5)
Statistical Analysis 1: Comparison: IFS Intervention Group vs Education Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, t-test, 2 sided — a priori threshold for statistical significance was <0.05; Mean Difference (Net) = 1.8, 95% CI 2-sided [0.5 to 3.1]

ADVERSE EVENTS:
Time Frame: All data was collected from the beiginning of the study in 2008 until study data collection was completed approximately 21 months after.
Arm/Group | IFS Intervention Group | Education Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

LIMITATIONS AND CAVEATS:
Participants declined participation due to long time frame. The attention given to the control group was less intense than the intervention group. There was greater attrition in the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No